CLINICAL TRIAL: NCT07044479
Title: A Clinical Study to Evaluate the Effects of Coffee and Tea on the Pharmacokinetics of Enlicitide in Healthy Adult Participants
Brief Title: A Clinical Study of How Coffee and Tea Affect Enlicitide in Healthy Volunteers (MK-0616-040)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0616-040; MK-0616-040 (Other: Merck)
Record Dates: First submitted 2025-06-26; First posted 2025-07-01 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Enlicitide Coffee Sequence 1 (Experimental): Participants will be randomized to receive enlicitide administered with water in period 1 and enlicitide with coffee in period 2.
  Interventions: Drug: Enlicitide
- Enlicitide Coffee Sequence 2 (Experimental): Participants will be randomized to receive enlicitide administered with coffee in period 1 and enlicitide with water in period 2.
  Interventions: Drug: Enlicitide
- Enlicitide Tea Sequence 1 (Experimental): Participants will be randomized to receive enlicitide administered with water in period 1 and enlicitide with tea in period 2.
  Interventions: Drug: Enlicitide
- Enlicitide Tea Sequence 2 (Experimental): Participants will be randomized to receive enlicitide administered with tea in period 1 and enlicitide with water in period 2.
  Interventions: Drug: Enlicitide

INTERVENTIONS:
Drug: Enlicitide — Single dose of enlicitide is administered orally on day 1 of each testing period
  Other Names: MK-0616; enlicitide decanoate

SUMMARY:
The goal of this study is to learn what happens to enlicitide in a person's body over time when enlicitide is taken at the same time as coffee or tea. Researchers will measure the amount of enlicitide in the blood when taken with coffee or tea compared with enlicitide taken with water.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health
* Is a non-smoker for at least 3 months prior to study entry
* Part 1 only: Consumes at least 1 cup of caffeinated coffee per day
* Part 2 only: Consumes at least 1 cup of caffeinated tea per day

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history or presence of clinically significant medical or psychiatric condition or disease
* History of gastrointestinal disease which might affect food and drug absorption, or has had gastric bypass or similar surgery.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Part 1-Coffee: Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Enlicitide | Predose and at designated time points up to 168 hours
  Blood samples will be collected to determine the AUC0-inf of enlicitide when administered with coffee
Part 1-Coffee: Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-last) of Enlicitide | Predose and at designated time points up to 168 hours
  Blood samples will be collected to determine the AUC from time 0 to the time of last quantifiable sample of enlicitide when administered with coffee
Part 1 -Coffee : Maximum Plasma Concentration (Cmax) of Enlicitide | Predose and at designated time points up to 168 hours
  Blood samples will be collected to determine the maximum observed drug concentration of enlicitide when administered with coffee
Part 2 -Tea: AUC0-last of Enlicitide | Predose and at designated time points up to 168 hours
  Blood samples will be collected to determine the AUC from time 0 to the time of last quantifiable sample of enlicitide when administered with tea
Part 2 - Tea: AUC0-Inf of Enlicitide | Predose and at designated time points up to 168 hours
  Blood samples will be collected to determine the AUC0-inf of enlicitide when administered with tea.
Part 2 -Tea: Cmax of Enlicitide | Predose and at designated time points up to 168 hours
  Blood samples will be collected to determine the maximum observed drug concentration of enlicitide when administered with tea

SECONDARY OUTCOMES:
Part 1 - Coffee: Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 7 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Part 2 - Tea: Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 7 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Part 1 - Coffee: Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 7 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.
Part 2 - Tea: Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 7 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion, Inc. ( Site 0001), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com